CLINICAL TRIAL: NCT04370678
Title: Changes in Preference for Surgery of Patients Signed up for Arthroscopic Procedures: COVID-19 Effect on Arthroscopic Patients in a University Hospital in Denmark
Brief Title: Changes in Preference for Surgery of Patients Signed up for Arthroscopic Procedures
Status: Completed | Type: Observational
Sponsor: Region Zealand (Other)
Responsible Party: Principal Investigator, Jesper Nielsen, Principal investigator, Region Zealand
Other Study IDs: ArthrocancellationSUH2020
Record Dates: First submitted 2020-04-24; First posted 2020-05-01 (Actual); Last update posted 2020-05-07 (Actual); Status verified 2020-05

CONDITIONS: Arthroscopy
Keywords: arthroscopy; shoulder impingement syndrome; Patient Preference; Covid-19; Public Health; Clinical Decision-Making
MeSH Terms: conditions — Shoulder Impingement Syndrome; Patient Preference; COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Change in preference to surgery under COVID-19 pandemic. — Under the COVID-19 pandemic all arthroscopic procedures were cancelled. We wished to describe if patients experienced a change in preference to surgery under this period.

SUMMARY:
This study describes the changes in preference to arthroscopic surgery in two orthopedics departments in Denmark under the COVID-19 pandemic.

DETAILED DESCRIPTION:
Background:

Covid-19 has impacted all aspects of society. In hospitals around the world focus has been on treating the deadly virus, and elective orthopedic surgical procedures has been postponed in Denmark, causing a stop for most arthroscopic procedures for months. It is established that certain conditions leading to arthroscopic orthopedic intervention has fluctuating symptoms symptoms and can have a favorable outcome on conservative treatment. Amongst these conditions who are also treated with non-surgical methods are subacromial decompression impingement[1][1], degenerative knee disease [2] and anterior cruciate ligament injuries[3]. An issue with further understanding the non-surgical effect on this patient group has beencould be reluctance to undergo conservative non-surgical treatment and opt for a surgical treatment. procedure. Because all elective surgery has been postponed in Denmark, and the following longer waiting period for surgery, this has created a unique opportunity to further investigate this patient category.

Aim of study: Investigate the impact of time on waiting list for surgery under COVID-19 pandemic on the preference for surgery in patients planned for arthroscopic surgery.

Discussion The current study will provide information on the change of preferences forto arthroscopic surgery in a patient population who are forced to wait for surgery for a longer period of time, with no possibility of seeking treatment in other hospitals.

ELIGIBILITY:
Inclusion Criteria:

* Patients planned for arthroscopic intervention in knee or shoulder.
* Patients seen by an orthopedic surgeon and planned for surgery before 13/3-20

Exclusion Criteria:

* Surgery performed in another hospital
* Death
* Emigration

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients planned for arthroscopic procedures at Zealand University Hospital in Køge in the time period 13-4-20 to 10-5-20.
Sampling Method: Non-Probability Sample
Enrollment: 79 (Actual)
Dates: Start 2020-04-17 (Actual); Primary Completion 2020-04-24 (Actual); Study Completion 2020-04-24 (Actual)

PRIMARY OUTCOMES:
Change in preference | 3 months
  change of preference for surgery during the waiting period for all planned arthroscopic procedures measured by questionnaire sent by letter asking if patients still want surgery yes or no. No other questions were asked.

SECONDARY OUTCOMES:
Change in preference between groups | 3 months
  difference in preference for surgery between the group of patients planned for arthroscopic procedure in the shoulder and patients planned for arthroscopic procedure in the knee measured by questionnaire sent by letter asking if patients still want surgery yes or no. No other questions were asked..

CONTACTS AND LOCATIONS:
Overall Officials: Jesper S Nielsen, MD, Principal Investigator — Zealand University Hospital, Køge
Locations (1):
- Zealand University Hospital, Køge, Region Sjælland, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Erratum: Treatments for Shoulder Impingement Syndrome: A PRISMA Systematic Review and Network Meta-Analysis: Erratum. Medicine (Baltimore). 2016 Jun 10;95(23):e96d5. doi: 10.1097/01.md.0000484495.36196.d5. eCollection 2016 Jun. PMID 31265590
- [Background] Brignardello-Petersen R, Guyatt GH, Buchbinder R, Poolman RW, Schandelmaier S, Chang Y, Sadeghirad B, Evaniew N, Vandvik PO. Knee arthroscopy versus conservative management in patients with degenerative knee disease: a systematic review. BMJ Open. 2017 May 11;7(5):e016114. doi: 10.1136/bmjopen-2017-016114. PMID 28495819
- [Background] Monk AP, Davies LJ, Hopewell S, Harris K, Beard DJ, Price AJ. Surgical versus conservative interventions for treating anterior cruciate ligament injuries. Cochrane Database Syst Rev. 2016 Apr 3;4(4):CD011166. doi: 10.1002/14651858.CD011166.pub2. PMID 27039329

DOCUMENTS (1):
  • Study Protocol (2020-04-24): https://cdn.clinicaltrials.gov/large-docs/78/NCT04370678/Prot_000.pdf